CLINICAL TRIAL: NCT05913856
Title: The Effectiveness of Oral Care With Chlorhexidine in Medical Intensive Care Unit:Ventilator-associated Pneumonia and Patient Outcomes
Brief Title: The Effectiveness of Oral Care With Chlorhexidine in Medical Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202106094RINC
Record Dates: First submitted 2023-06-04; First posted 2023-06-22 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-08

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Saline Solution; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorhexidine group (Experimental): Applying 0.12% chlorhexidine mouthwash for oral care thrice daily.
  Interventions: Other: Chlorhexidine
- Normal saline group (Active Comparator): Applying normal saline for oral care thrice daily.
  Interventions: Other: Normal saline

INTERVENTIONS:
Other: Normal saline — Normal saline will be applied to irregate the oral cavity after the swabing of the surface of patients' teeth and oral cavity by a sponge swab by the primary care nurse in the MICU.
  Arms: Normal saline group
Other: Chlorhexidine — 15ml of 0.12% chlorhexidine will be applied to irregate the oral cavity after the swabing of the surface of patients' teeth and oral cavity by a sponge swab by the primary care nurse in the MICU.
  Arms: Chlorhexidine group

SUMMARY:
Oral care with chlorhexidine was used to be considered an effective way to prevent ventilator-associated pneumonia (VAP). However, recent evidence revealed that oral care with chlorhexidine may associate with higher mortality and increasing risks of acute respiratory distress syndrome due to the aspiration of chlorhexidine. In addition, the majority of relevant studies in the past have only focused on cardiothoracic intensive care unit (ICU) or post-operation patients. Thus, whether this is effective and safe for medical ICU patients remains unclear.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is one of the most common hospital-acquired infections in the ICU, associated with an increased hospital stay, increased cost of treatment, prolonged ventilator days, and increased morbidity and mortality rates (Divatia et al, 2019). The overall incidence of VAP was around 12% in Asia and nearly 8% in Taiwan in the past 30 years (Bonell et al, 2019), with a mortality rate that may exceed 45% for those receiving mechanical ventilation (Feng et al, 2019). Therefore, the prevention of VAP is a key part of managing patients undergoing mechanical ventilation.

Oral decolonization by mouthwash using a chlorhexidine-contained solution was suggested by accumulated evidence in preventing VAP (Dai et al, 2022). However, controversial opinions existed from a few different points of view. First of all, Klompas et al (2014) conducted a meta-analysis that showed the effectiveness of chlorhexidine (CHG) oral care in preventing VAP was limited only to cardiac surgery patients (Klomopas et al, 2014). Second, recent evidence showed a possibility of unfavored outcomes related to the use of CHG mouthwash by increased mortality either in the ICU (Price et al, 2014) or the general ward (Deschepper et al, 2018). Last but not least, the subjectiveness of the diagnostic criteria of VAP had led to the discussion on the credibility of the outcome in relevant studies (Skrupky et al, 2016). Therefore, the US Centers for Disease Control and the National Healthcare Safety Network have proposed alternative diagnostic criteria for the ventilator-associated event (VAE) as alternation (Peña-López et al, 2022).

The objective of this study was to examine the effectiveness of oral care with 0.12% CHG in MICU patients for the prevention of ventilator-associated events.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 20 years old
* admitted to MICU
* an oral endotracheal tube inserted under mechanically ventilated

Exclusion Criteria:

* an endotracheal tube inserted over 24 hours before enrollment
* intubated because of trauma, burn, operation, or neurological disease
* already suffered from oral ulcers before intubation
* known history of allergic reaction to CHG
* use of ECMO

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of ventilator-associated event within ICU admission | Will be surveyed retrospectively through study completion within 3 months
  The US CDC has proposed an objective diagnostic criteria to identify adverse events during mechanical ventilation, which comprises three levels: ventilator-associated condition (VAC), infection-related ventilator-associated condition (IVAC), and possible ventilator-associated pneumonia (PVAP).

SECONDARY OUTCOMES:
ICU length of stay | Will be surveyed retrospectively through study completion within 3 months
  The total duration of the patient's ICU stay (days).
Hospital length of stay | Will be surveyed retrospectively through study completion within 3 months
  The total duration of the patient's hospital stay (days).
ICU mortality | Will be surveyed retrospectively through study completion within 3 months
  Whether the patient has died during their stay in the ICU
Hospital mortality | Will be surveyed retrospectively through study completion within 3 months
  Whether the patient has died during their stay in the hospital
Changes in the oral health status evaluated by the Beck Oral Assessment Scale | The surveys will be conducted within 24 hours of patient enrollment, within the fourth day after the patient is intubated, and within the 1 day following extubation.
  The status of oral health will be evaluated using the Beck Oral Assessment Scale by the researcher, which provides a comprehensive evaluation of oral health by assessing various parameters such as lips, tongue, gums, and teeth.
Changes in the oral health status evaluated by the Mucosal-Plaque Score | The surveys will be conducted within 24 hours of patient enrollment, within the fourth day after the patient is intubated, and within the 1 day following extubation.
  The status of oral health will be evaluated using the Mucosal-Plaque Score by the researcher, which focuses specifically on assessing the presence and extent of mucosal inflammation and plaque accumulation in the oral cavity.
Incidence of Ventilator-Associated Pneumonia | From the date of intubation until the first occurrence of extubation or in-ICU death, whichever occurs first, assessed up to 28 days.
  Ventilator-associated pneumonia (VAP) will be included as an additional secondary outcome. Diagnosis of VAP will follow the 2016 Infectious Diseases Society of America (IDSA) and American Thoracic Society (ATS) clinical practice guidelines.
  A case of VAP is defined by the presence of a new or progressive pulmonary infiltrate on chest radiograph, plus at least two of the following clinical features:
  Fever >38°C or hypothermia <36°C,leukocytosis (>12,000/μL) or leukopenia (<4,000/μL), or purulent tracheal secretions.
  Chart reviews will be conducted in a two-step process: (1) initial screening by trained research staff based on clinical documentation (excluding radiographic findings), and (2) blinded interpretation of chest X-rays by a physician reviewer. The diagnostic window for VAP will be based on the temporal cluster of clinical signs, typically within ±48 hours. The outcome will be reported as the number of VAP cases per group, and if data permits, as incidence per 1,000 ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chen Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National taiwan university hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No